CLINICAL TRIAL: NCT03127917
Title: Impact of Reduced Arterial Stiffness on Peripheral Vascular Function and Mobility
Brief Title: Effect of L-Citrulline on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Joaquin U Gonzales, PhD, Associate Professor, Texas Tech University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 15BGIA22710012
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Citrulline; Blood Flow; Aging
Keywords: Gait Speed; Cognitive Function
MeSH Terms: interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind research study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CitrullinePlacebo (Experimental): Subjects allocated to the CitrullinePlacebo study arm received L-citrulline first, followed by placebo.
  Interventions: Dietary Supplement: L-citrulline; Other: Placebo
- PlaceboCitrulline (Experimental): Subjects allocated to the PlaceboCitrulline study arm received placebo first, followed by L-citrulline.
  Interventions: Dietary Supplement: L-citrulline; Other: Placebo

INTERVENTIONS:
Dietary Supplement: L-citrulline — L-citrulline capsules given at 6 g/day
Other: Placebo — Maltodextrin capsules given as placebo

SUMMARY:
The objective of this project is to determine the importance of peripheral vascular function on gait performance in older adults.

DETAILED DESCRIPTION:
This project employed a placebo controlled, double-blind, crossover trial. Participants were randomized to oral L-citrulline (6 g/day) or placebo (maltodextrin) for 14 days, and switched to the other treatment for another 14 days after washout. Peripheral vascular function was assessed under conditions of rest, leg exercise, and cognitive engagement. Gait performance was assessed using clinical walking tests.

ELIGIBILITY:
Inclusion Criteria:

* older adults
* women and men
* aged 60-79 yrs
* must be able to swallow capsules
* fully mobile without assistive walking devices

Exclusion Criteria:

* have physician diagnosed cardiovascular, pulmonary, or metabolic disease
* are current smokers
* currently taking medications affecting cardiovascular function
* have high blood pressure (>159/99 mmHG)
* have high fasting blood glucose (>110 mg/dL)
* are considered obese (body mass index ≥ 30 kg/m2)
* have orthopaedic limitations that limit walking ability
* have pacemaker or other metal objects in their body

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Blood Flow | baseline and 2 weeks for L-citrulline and placebo
  Femoral blood flow during leg exercise and carotid blood flow during mental activity measured using Doppler ultrasound. Blood-oxygen-level dependent contrast imaging of the brain using functional magnetic resonance imaging (fMRI) during cognitive functioning.

SECONDARY OUTCOMES:
Gait Performance | baseline and 2 weeks for L-citrulline and placebo
  Usual and fast walking speeds measured during short (7m) and long (400m) distances.

IPD SHARING:
Plan to Share IPD: Yes
Raw data for outcome variables will be made available on the online general repository "figshare" within 12 months of funding end date.
Time Frame: Within 12 months of funding end date.
Access Criteria: Use these two URL's to access different data sets and associated published work.
  https://figshare.com/s/1b382cb5e788663047e7 https://figshare.com/s/c45b46f67391b140f774
URL: https://figshare.com/s/c45b46f67391b140f774